CLINICAL TRIAL: NCT03112304
Title: Child STEPS for Youth Mental Health in Maine: Sustainability of MATCH in the Public Sector
Brief Title: Child STEPS for Youth Mental Health in Maine Sustainability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, John Weisz, Primary Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H030711
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Anxiety; Depression; Trauma; Behavior Problems
Keywords: children; youth; adolescents; anxiety; depression; trauma; behavior problems; evidence-based treatments; manualized; cognitive-behavioral therapy; mental health
MeSH Terms: conditions — Anxiety Disorders; Depression; Wounds and Injuries; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MATCH-ADTC Wave 1 (Experimental): Wave 1 clinicians received MATCH training at the beginning of the project and used MATCH to treat participating children from their clinic for two years, with weekly case consultation from MATCH experts who were part of the study team, and then received consultation from their own clinic supervisors who had been trained as MATCH Associate Consultants (ACs), supported by the TRAC system.
  Interventions: Behavioral: MATCH-ADTC; Other: TRAC
- MATCH-ADTC Wave 2 (Experimental): Wave 2 clinicians provided treatment as usual (e.g., usual care) with the children they treated during the initial two years of the project. Afterwards, they trained in MATCH and used it to treat children in their clinics with weekly case consultation from our study team of MATCH experts, supported by the TRAC system.
  Interventions: Behavioral: MATCH-ADTC; Other: TRAC

INTERVENTIONS:
Behavioral: MATCH-ADTC — MATCH - ADTC (Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems; Chorpita & Weisz, 2009) is a psychosocial intervention designed to treat children with multiple disorders and problems encompassing anxiety, depression, post-traumatic stress, and disruptive conduct, including the conduct problems associated with ADHD. It is recommended for children aged 6-15. MATCH is composed of 33 modules-i.e., specific treatment procedures derived from decades of research on EBTs. The various modules can be organized and sequenced flexibly to tailor treatment to each child's characteristics and needs.
  Other Names: MATCH
Other: TRAC — TRAC (Treatment Response Assessment for Children) is a web-based system that provides weekly monitoring of the MATCH modules used and the child's response to treatment. Child's response to treatment is based on caregiver and child reports of (a) changes in problem severity on the standardized Brief Problem Checklist, and (b) changes in severity of the top treatment concerns identified by youths and caregivers. At the end of treatment, TRAC provides a complete record of modules used, and child treatment response, across all the weeks of treatment, as illustrated in the "client dashboard."

SUMMARY:
The overarching goal of this project is to study the sustainability of MATCH-ADTC within community mental health clinics, to learn what is needed for evidence-based practices (EBPs) to take root and thrive within a public system.

DETAILED DESCRIPTION:
In this project, the investigators are randomizing children to Wave 1 (previously MATCH trained) or Wave 2 (newly MATCH trained) and using a clinical monitoring system (TRAC) to measure youth outcomes over time. Participating therapists receive weekly MATCH consultation provided by the Judge Baker Children's Center/Harvard University research team or by Maine clinic supervisors who are MATCH Associate Consultants. The investigators are also developing and testing new low-cost measures of MATCH treatment and consultation fidelity to explore the feasibility of more sustainable measures of MATCH adherence. Study data will be used to answer questions about the sustainability of MATCH in the public sector.

ELIGIBILITY:
Inclusion Criteria:

* 6 - 15 year old child and their caregivers
* seeking services at community mental health clinics
* primary problem or disorder related to anxiety, traumatic stress, depression, or conduct problems, or any combination of the four problems

Exclusion Criteria:

* child is younger than 6 years or older than 15 years on the day of the phone screen.
* child has attempted suicide within the past year.
* Schizophrenic spectrum disorder (including MDD with psychotic features)
* Autism or another Pervasive Developmental Disorder (E.g., PDD NOS, Asperger's Disorder, Child Disintegration Disorder, Rett's Disorder)
* Anorexia Nervosa
* Bulimia Nervosa
* Mental Retardation
* no relevant T-scores validate target disorders
* ADHD identified as primary reason for seeking treatment at phone screen
* child's medication has not been regulated for one month or longer

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Brief Problem Checklist (BPC) | Change over time from Day 1 to Day 242 (end of treatment)
Top Problems Assessment (TPA) | Change over time from Day 1 to Day 534 (18 month follow-up)

SECONDARY OUTCOMES:
Youth Self-Report and Child Behavior Checklist | Change over time from Day 1 to Day 534 (18 month follow-up)
Therapeutic Alliance Scale for Children (TASC) | Change over time from Day 1 to Day 267(end of treatment)
Client Satisfaction Questionnaire- 8 (CSQ-8 ) | Change over time from Day 1 to Day 267(end of treatment)
Youth Satisfaction Questionnaire-8 (YSQ-8) | Change over time from Day 1 to Day 267(end of treatment)
Therapist Satisfaction Inventory (TSI) | Change over time from Day 1 to Day 267(end of treatment)
Evidence-Based Practice Attitudes Scale (EBPAS) | Change over time from Day 1 to Day 267(end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: John R Weisz, PhD, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Chorpita, B.F., & Weisz, J.R. (2009). Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems (MATCH-ADTC). Satellite Beach, FL: PracticeWise, LLC.